CLINICAL TRIAL: NCT01233492
Title: A Cancer Research UK Pharmacokinetic Study of BPA in Patients With High Grade Glioma to Optimize Uptake Parameters for Clinical Trials of BNCT
Brief Title: Boron Phenylalanine With or Without Mannitol in Treating Patients With Glioblastoma Multiforme
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Cancer Research UK (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000687653; CRUK-PH1/093; EUDRACT-2004-002413-37
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Mannitol

INTERVENTIONS:
Drug: boron phenylalanine
Drug: mannitol
Other: biologic sample preservation procedure
Radiation: radiation therapy treatment planning/simulation

SUMMARY:
RATIONALE: Giving boron phenylalanine in different ways and measuring it in tissue in patients with glioblastoma multiforme may help in planning better radiation therapy, such as boron neutron capture therapy, for patients in the future.

PURPOSE: This phase I trial is studying the side effects, best dose boron phenylalanine, and best way of giving it with or without mannitol in treating patients with glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the optimal way to deliver boron phenylalanine (BPA) with or without mannitol in terms of route (intravenous vs intraarterial), blood-brain barrier disruption, and dose for use in subsequent therapeutic trials of boron neutron capture therapy (BNCT) in patients with high-grade glioma.
* To evaluate the toxicity profile of BPA administered intravenously or intra-arterially.
* To evaluate the pharmacokinetic behavior of BPA using samples of blood, urine, tumor tissue, normal brain tissue, extracellular fluid, and cerebrospinal fluid.

Secondary

* To produce indicative treatment plans using BPA administered either intravenously or intra-arterially with or without mannitol to support the design of combination studies using BPA and thermal neutrons for BNCT.

Tertiary

* To evaluate the micro-distribution of boron resulting from the different routes of administration using secondary ion mass spectroscopy (SIMS).
* To store surplus tissues removed during the trial for possible future studies.

OUTLINE: This is a dose-escalation study.

* Stage 1 (Route and Blood Brain Barrier Disruption [BBBD]): Patients receive one dose of boron phenylalanine intravenously (IV) or intra-arterially (IA) over 2 hours. Some patients may receive mannitol IA over 30 seconds before receiving boron phenylalanine. Patients then undergo planned biopsy of the tumor. Some patients may then undergo immediate surgical debulking of the tumor.

Boron distribution data is analyzed to determine the optimal administration schedule. Patients in stage 2 receives boron phenylalanine via the optimal route established in stage 1. If addition of mannitol is found to be beneficial, then mannitol is used in stage 2

* Stage 2 (Dose-escalation): Patients receive 1 or 2 doses of boron phenylalanine IV or IA (as determined in stage 1) over 2 hours on day 1. Patients may also receive mannitol IA as in stage 1.

Tumor tissue, normal brain tissue, and cerebrospinal fluid are collected during biopsy and/or surgery. Some patients undergo blood, urine, extracellular fluid sample collection periodically for pharmacokinetic studies. Tumor tissue will be stored for future studies.

After completion of study treatment, patients are followed for 7 days and then once a month.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Radiologically and clinically suspected solitary glioblastoma multiforme

  * High-grade disease
* Agreed to undergo stereotactic biopsy as part of routine diagnostic work-up

PATIENT CHARACTERISTICS:

* WHO performance status 0-2 (0-1 for patients ≥ 65 years old)
* Life expectancy > 4 months
* Hemoglobin ≥ 9.0 g/dL
* Neutrophil count ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Serum bilirubin ≤ 1.5 times upper normal of limit (ULN)
* AST ≤ 1.5 times ULN
* Uncorrected EDTA-Isotope creatinine clearance ≥ 40 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use two forms of effective contraception 4 weeks prior to, during, and for 6 months after completion of study therapy
* Able to cooperate with procedures and follow-up
* Not at high risk of complications from blood-brain barrier disruption with mannitol on pre-treatment CT scan (an open quadrigeminal plate cistern, absence of dilatation of the contralateral frontal horn, and absence of uncal herniation)
* No history of uncontrolled seizures
* No phenylketonuria
* No current or previous malignancies at sites other than the brain, except for adequately treated cone-biopsied carcinoma in-situ of the uterine cervix or basal cell or squamous cell carcinoma of the skin
* Not at high medical risk due to nonmalignant systemic disease, including active uncontrolled infection
* No known hepatitis B, hepatitis C, or HIV positivity by serology
* No concurrent congestive heart failure, history of NYHA class III-IV cardiac disease, history of myocardial infarction or active ischemic heart disease within the past year, or history of cardiac arrhythmia or thromboembolic disease
* No other condition that, in the investigator's opinion, would not make the patient a good candidate for the clinical trial

PRIOR CONCURRENT THERAPY:

* At least 12 hours since prior and no concurrent steroids
* At least 48 hours since prior phenylalanine-containing drinks (e.g., colas)
* At least 48 hours since prior excessive consumption of phenylalanine-containing foods, including any of the following:

  * Low phenylalanine content (e.g., fruit juice, fruits [except bananas], vegetables, and low-protein breads and pastas
  * Medium phenylalanine content (e.g., corn, bread, french fries, potatoes, peas, rice, and regular pasta)
  * High phenylalanine content (e.g., refried beans, chicken, nuts, hamburgers, peanuts, cheese, eggs, pork chops, steak, bananas, and milk)
* At least 4 weeks since prior major thoracic and/or abdominal surgery and recovered
* No prior cranial radiotherapy
* No prior endocrine therapy, immunotherapy, or chemotherapy for the brain tumor
* No other concurrent anticancer therapy or investigational drugs

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2007-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Optimal dose of boron phenylalanine (BPA)
Causality of each adverse event to BPA and grading severity according to NCI CTCAE Version 3.0
Pharmacokinetic (PK) parameters used to construct a PK model with the aim of being able to predict boron up-take by tumor and normal brain tissue

SECONDARY OUTCOMES:
Change in mean dose to the planning target volume of greater than 15%, for a constant maximum and mean dose to normal tissue in any treatment cohort of the study
Change in the intra-nuclear percentage of 10B atoms in any cohort of the study of greater than 20%
Establishment of a repository of samples including serum and tumor tissue for future studies using techniques such as proteomics and DNA array

CONTACTS AND LOCATIONS:
Overall Officials: Garth Cruickshank, Principal Investigator — University Hospital Birmingham
Locations (2):
- United Kingdom (2):
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - Cancer Research UK Clinical Trials Unit - Birmingham, Birmingham, England